CLINICAL TRIAL: NCT03073603
Title: Discontinuation of Disease Modifying Therapies (DMTs) in Multiple Sclerosis (MS)
Acronym: DISCOMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Multiple Sclerosis Society (Other); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-2388
Record Dates: First submitted 2017-01-18; First posted 2017-03-08 (Actual); Results first posted 2022-10-06 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug Continuation Arm (Active Comparator): Participants who remain on their current Disease Modifying Therapies (DMTs) without any changes. DMTs include ~14 formulations/doses of drugs approved in the US by the FDA that alter the natural history of the disease.
  Interventions: Drug: Standard of Care
- Drug Discontinuation Arm (Experimental): Participants who will discontinue their Disease Modifying Therapies (DMTs). No other changes to their treatment occur. DMTs include ~14 formulations/doses of drugs approved in the US by the FDA that alter the natural history of the disease.
  Interventions: Drug: Discontinuation of disease modifying therapy

INTERVENTIONS:
Drug: Discontinuation of disease modifying therapy — Participants who will discontinue their current MS drug. No other changes to their treatment occur.
  Arms: Drug Discontinuation Arm
Drug: Standard of Care — Participants who remain on their current Disease Modifying Therapies (DMTs) without any changes. DMTs include ~14 formulations/doses of drugs approved in the US by the FDA that alter the natural history of the disease.
  Arms: Drug Continuation Arm

SUMMARY:
Natural history research in Multiple Sclerosis (MS) suggests that risk of relapses and new Magnetic Resonance Imaging (MRI) changes diminish significantly as people age, especially in MS patients 55 or older. Thus, the need to continue MS medicines that reduce relapses and new MRI lesions may also decrease as people age, especially in those who have not had relapses or MRI scan changes for prolonged times. This study plans to learn more about the safety of stopping MS medication in this population, as compared to continuing on the medication.

DETAILED DESCRIPTION:
Participants will be randomized (1:1) to one of two groups. One group will stay on their current MS medication (Continue group), and one group will discontinue their medication (Discontinue group). They will also have some extra assessments done at their regular routine MS clinic appointment and every 6 months for the next 18-24 months. The following items will be done in addition to any assessments or procedures they are already having done as part of their clinical care:

* Questionnaires about the participant's quality of life including questions about health, mood, thinking, and social life
* Questionnaires about the participant's MS symptoms
* Test of the participant's attention, concentration, and thinking
* Test of the participant's physical symptoms
* In addition to any MRIs the participants may get as part of their routine care, they will also have an MRI 6 months from their enrollment into the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either Relapsing-remitting MS (RRMS), Secondary progressive MS (SPMS), or Primary progressive MS (PPMS) by McDonald 2010 criteria.
* Patients defined by subtype based on 2013 updated phenotypic criteria.
* Progression of MS defined by the local PI either:

  * prospectively with an EDSS change of at least 1.0 points over the last two years, or
  * retrospectively, with any significant change in motor function over at least one year, unrelated to relapse.
* 55 years of age or older at time of randomization;
* No evidence of recent new inflammatory disease activity (inactive by the Lublin criteria16) with no new relapse for at least five years and no new MRI lesion for at least three years
* Using any of the FDA-approved MS DMTs (to include:

  * interferon β-1a,
  * interferon β-1b,
  * glatiramer acetate,
  * natalizumab,
  * fingolimod,
  * dimethyl fumarate,
  * ocrelizumab, or
  * teriflunomide; continuously for no less than 5 years.
* Taking most recent DMT continuously* for no less than two years.
* Willing to be randomized per this protocol; each patient will be questioned as to their willingness to stay in the trial regardless of the group to which group they are randomized.
* Willing to follow the protocol
* Able to undergo a brain MRI without anesthesia

  * Continuously will be defined as no less than 75% of all prescribed doses, with no time of greater than four weeks from last intended dose to have missed a dose (8 weeks for natalizumab, i.e. one missed dose).

Exclusion Criteria:

* Any MS relapse in the last five years, as determined at the screen visit by the PI
* Any new or definitely enlarging T2/FLAIR lesion or new gadolinium-enhancing lesion within the past three years (at least two scans separated by at least three years must be reviewed) on brain or spine MRI scan. Lesions must be 3mm or larger to be exclusionary.
* Significant (as defined by the PI) intolerance of presently-used DMT
* More than two courses of acute, systemic (IV or oral) steroids in the last 5 years or any use within the last year. Course is defined as three or more days continuously, and not to exceed 14 days. No use of chronic, systemic steroids, defined as 15 or more days, in the last 5 years. Any use of steroids to treat MS relapse, possible relapse, or pseudo-relapse in the last 5 years.

  * Use of inhaled or topical steroids are not an exclusion criteria.
  * Use of oral steroids for no greater than 14 days given for a non-MS condition is not exclusionary.
* Prior use of the following in the past 5 years:

  * alemtuzumab,
  * mitoxantrone,
  * cyclophosphamide,
  * methotrexate,
  * cyclosporine,
  * rituximab,
  * siponimod, or
  * cladribine
* Prior use of any experimental agent used as a DMT for MS in the last five years
* Other significant medical or psychiatric illness, if uncontrolled. Examples:

  * uncontrolled hypertension,
  * uncontrolled diabetes,
  * uncontrolled asthma, or
  * uncontrolled depression
* Cancers other than basal cell skin cancers within the last 5 years
* Unable to give informed consent or follow the protocol
* Unable to undergo brain MRI
* Unwilling to be randomized per this protocol
* History of other chronic neurological illnesses that might mimic MS with chronic or intermittent symptoms (i.e. ALS, myasthenia gravis, chronic neuropathy, etc.)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Corboy, MD, Principal Investigator — University of Colorado, Denver
Locations (19):
- United States (19):
  - University of Southern California, Los Angeles, California
  - University of Colorado Denver - Anschutz Medical Campus, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University St. Louis, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Mt. Sinai University, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Swedish Health Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corboy JR, Fox RJ, Kister I, Cutter GR, Morgan CJ, Seale R, Engebretson E, Gustafson T, Miller AE; DISCOMS investigators. Risk of new disease activity in patients with multiple sclerosis who continue or discontinue disease-modifying therapies (DISCOMS): a multicentre, randomised, single-blind, phase 4, non-inferiority trial. Lancet Neurol. 2023 Jul;22(7):568-577. doi: 10.1016/S1474-4422(23)00154-0. PMID 37353277
- [Derived] Hartung HP, Meuth SG, Miller DM, Comi G. Stopping disease-modifying therapy in relapsing and progressive multiple sclerosis. Curr Opin Neurol. 2021 Aug 1;34(4):598-603. doi: 10.1097/WCO.0000000000000960. PMID 33990101
- [Derived] McGinley MP, Cola PA, Fox RJ, Cohen JA, Corboy JJ, Miller D. Perspectives of individuals with multiple sclerosis on discontinuation of disease-modifying therapies. Mult Scler. 2020 Oct;26(12):1581-1589. doi: 10.1177/1352458519867314. Epub 2019 Aug 1. PMID 31368401

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Started | 128 | 131
Completed | 106 | 123
Not Completed | 22 | 8
Not completed — Noncompliance | 3 | 1
Not completed — Adverse Event | 5 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Required treatment not allowed by protocol | 1 | 0
Not completed — Financial or insurance-related | 8 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Discontinued DMT | 4 | 0
Not completed — Restarted DMT | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm | Total
Number analyzed (Participants) | 128 | 131 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (5.2) | 63.1 (4.9) | 63.0 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 109 | 216
  Male | 21 | 22 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 12 | 11 | 23
  Hispanic | 1 | 1 | 2
  White | 112 | 119 | 231
  Other | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 128 | 131 | 259
MS Phenotype [Count of Participants; unit: Participants]
  Primary Progressive | 2 | 6 | 8
  Secondary Progressive | 18 | 17 | 35
  Relapsing-Remitting | 108 | 108 | 216
Time since first onset of symptoms related to MS [Mean (Standard Deviation); unit: years] | 20.9 (10.4) | 23.4 (10.5) | 22.2 (10.5)
Time since last documented relapse [Mean (Standard Deviation); unit: years] | 13.2 (6.2) | 14.5 (7.4) | 13.9 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Developing a New MS Relapse and/or MRI Brain Lesion Over the Course of the Study Duration
Description: The outcome is the proportion of participants in each group developing a new MS relapse and/or MRI brain lesion over the course of the study duration. Count of Participants with either a new MS relapse and/or a new brain MRI lesion is reported.
Time Frame: 18-24 months, based on time of enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 128 | 131
Participants | 6 | 16
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; We tested the null hypothesis of inferiority with the proportion of disease events (i.e., new MS relapse and/or MRI brain lesion) for the drug discontinuation group being 8% greater than the proportion for the drug continuation group under the alternative that the two rates are equal; Test type: Non-Inferiority — We performed a non-inferiority test for the proportions of the drug continuation and drug discontinuation arms experiencing a new MS relapse and/or MRI Brain Lesion over the course of the study duration. The non-inferiority margin used was 8%; p = 0.521, Exact binomial test; Exact binomial test for difference in two proportions; Difference in proportion = 0.0753, 95% CI 2-sided [0.0063 to 0.1500]

2. Secondary Outcome: Number With Disability Progression Confirmed at 6 Months Using the Expanded Disability Status Scale (EDSS)
Description: The EDSS is a neurological examination performed by a blinded rater. This assessment is collected at each study visit. Increase in the EDSS score shows disease activity or progression, and must be observed six months later to be confirmed. Whether a confirmed change is significant depends on the subject's EDSS at baseline: for those with a baseline EDSS of 5.5 points or fewer, the increase must be at least one point to be significant; for those with a baseline EDSS of 6.0 points or greater, a change of at least 0.5 points is considered significant. We will calculate the percentage in each group of those who had a significant change at anytime during the follow-up period, which was then confirmed at 6 months later.
Time Frame: Baseline, then every 6 months for up to a maximum of 24 months, based on time of enrollment.
Population: Three subjects (2 in drug continuation arm and 1 in drug discontinuation arm) did not have a baseline EDSS recorded, so change in EDSS could not be assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 126 | 130
Participants | 14 | 16
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.766, Chi-squared

3. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Upper Extremity Function
Description: The Neuro-QOL Adult PRO short form measures are collected to evaluate self-reported overall quality of life and functioning in patients with a variety of neurological conditions including MS. The Neuro-Qol short form scales consist of 5-9 single scale item scales. Raw scores are then converted to a standardized score with mean 50 and standard deviation 10. The Neuro-QoL short forms used in this study with higher scores representing better outcomes are: Upper Extremity Function, Lower Extremity Function, Cognitive -- General Concerns, Cognitive -- Executive Function, Communication, Positive Affect and Well-Being, Satisfaction with Social Roles and Activities, and Ability to Participate in Social Roles and Activities. The short forms used with lower scores representing better outcomes are: Fatigue, Sleep Disturbance, Anxiety, Depression, and Emotional-Behavioral Dyscontrol.
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 109 | 113
units on a scale | -1.1 (6.2) | -0.6 (5.8)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.604, t-test, 2 sided

4. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Lower Extremity Function
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 108 | 113
units on a scale | -0.2 (5.5) | -1.1 (5)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.198, t-test, 2 sided

5. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Fatigue
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 109 | 113
units on a scale | -0.1 (6.2) | -0.9 (6.8)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.354, t-test, 2 sided

6. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Sleep Disturbance
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 108 | 113
units on a scale | -0.3 (5.6) | -0.5 (5.7)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.831, t-test, 2 sided

7. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- General Concerns
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 109 | 112
units on a scale | 0.6 (5.6) | 1.5 (6.4)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.252, t-test, 2 sided

8. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Executive Function
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 105 | 112
units on a scale | 0.3 (6.3) | 0.3 (6.2)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.983, t-test, 2 sided

9. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Communication
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 105 | 109
units on a scale | 0.1 (2.2) | -0.4 (3)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.155, t-test, 2 sided

10. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Anxiety
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 108 | 113
units on a scale | 0.2 (6) | 0.4 (6.2)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.748, t-test, 2 sided

11. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Depression
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 108 | 112
units on a scale | 0.9 (4.9) | 1.1 (5.5)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.773, t-test, 2 sided

12. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Positive Affect and Well-Being
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 108 | 113
units on a scale | 0 (6.3) | -1.2 (8.2)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.224, t-test, 2 sided

13. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Emotional-Behavioral Dyscontrol
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 109 | 112
units on a scale | -0.2 (7.8) | -0.3 (7.2)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.962, t-test, 2 sided

14. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Satisfaction With Social Roles and Activities
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 105 | 113
units on a scale | 1.7 (6.9) | -0.7 (5.7)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.005, t-test, 2 sided

15. Secondary Outcome: Change in Neuro-QoL (Quality of Life) Short Form Scores -- Ability to Participate in Social Roles and Activities
Description: as for outcome 3
Time Frame: Baseline, 18-24 Months, based on time of enrollment
Population: Subjects missing Neuro-QOL at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 105 | 112
units on a scale | -2.8 (10) | -1.6 (11)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.406, t-test, 2 sided

16. Secondary Outcome: Change in SymptoMScreen Composite Score (SymptoMScreen - Overall Symptom Severity).
Description: SymptoMScreen will be collected to assess overall symptom severity. Participants self-report across multiple neurological domains (mobility, hand function, spasticity, pain, sensory, bladder, fatigue, vision, dizziness, cognition, depression, and anxiety). This scale is a single page, validated measure that allows for quick assessment of multiple symptoms. Single item scores are rated as 0-6 with higher numbers representing increased limitations and symptom severity. Composite score is calculated by summing the single item scores with total score ranges from 0 to 72.
Time Frame: Baseline, then every 6 months for up to a maximum of 24 months, based on time of enrollment. The change between baseline and Month 18-24 is reported.
Population: Subjects missing SymptoMScreen at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 113 | 118
units on a scale | 0 (0.5) | 0 (0.5)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.348, t-test, 2 sided

17. Secondary Outcome: Change in Patient-Determined Disease Steps (PDDS - Disability).
Description: Patient-Determined Disease Steps will be collected to assess changes in disability from the patient's perspective. This outcome measure is a single question. The scores range from 0 to 8, and a participant with a low score has less perceived disability than a participant with a higher score.
Time Frame: as for outcome 16
Population: Subjects missing PDDS at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 107 | 115
units on a scale | 0 (1.1) | 0.3 (1.1)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.086, t-test, 2 sided

18. Secondary Outcome: Change in Symbol Digit Modalities Test (SDMT - Cognition).
Description: The SDMT measures patient attention, concentration, and speed of information processing and has been validated for discriminating patients from controls. Possible scores range from 0 to 110, with higher scores indicating a better outcome.
Time Frame: as for outcome 16
Population: Subjects missing SDMT at either baseline or at Month 18-24 were excluded from this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 108 | 112
units on a scale | 2.5 (9.6) | 1.8 (8.8)
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.575, t-test, 2 sided

19. Secondary Outcome: Evaluation of the Patient's Quality of Life Using the MSIS-29 Scale -- Physical Impact
Description: The Multiple Sclerosis Impact Scale (MSIS-29) will be collected to assess changes in quality of life from the patient's perspective. The MSIS has 29 questions. Each question asks the participant to rank how impacted they are in a certain aspect of their life. The options are 1 through 4. 1 indicates not at all impacted while 4 indicates extremely impacted. The lower the final score, the less impacted the participant is overall. Scores on the physical impact scale range from 20-80 and from 9-36 on the psychological impact scale. We will compare the proportion in each group who have had a change of 7.5 points or more (considered a clinically meaningful change).
Time Frame: as for outcome 16
Population: Subjects missing MSIS-29 at either baseline or at Month 18-24 were excluded from this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 113 | 117
Participants | 41 | 45
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.733, Chi-squared

20. Secondary Outcome: Evaluation of the Patient's Quality of Life Using the MSIS-29 Scale -- Psychological Impact
Description: as for outcome 19
Time Frame: as for outcome 16
Population: Subjects missing MSIS-29 at either baseline or at Month 18-24 were excluded from this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 113 | 117
Participants | 44 | 43
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.733, Chi-squared

21. Other Pre Specified Outcome: Total Number of New T2 Lesions on MRI
Description: MRIs will be reviewed to determine the total number of new T2 lesions that develop for each subject over the course of the study. Lesion counts will be performed by the central MRI facility.
Time Frame: Baseline, then every 6 months for 2 years with one exception at 18 months.
Measure: Median (Full Range); unit: lesions
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
Number analyzed (Participants) | 128 | 131
lesions | 0 [0 to 2] | 0 [0 to 5]
Statistical Analysis 1: Comparison: Drug Continuation Arm vs Drug Discontinuation Arm; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (24 months)
Description: All SAEs are reported in the table of Serious Adverse Events.
  Other adverse events exceeding a frequency threshold of 5% are reported. Additionally, AEs were classified as being unrelated to treatment, unlikely to be related to treatment, possibly (> 50% likelihood) related to treatment, probably related to treatment, or definitely related to treatment. Any AEs deemed probably or definitely related to treatment are reported, even if they did not exceed the 5% threshold.
Arm/Group | Drug Continuation Arm | Drug Discontinuation Arm
All-Cause Mortality (participants affected / at risk) | 1/128 | 2/131
Serious Adverse Events (participants affected / at risk) | 1/128 | 1/131
Other Adverse Events (participants affected / at risk) | 66/128 | 70/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Continuation Arm (N=128) | Drug Discontinuation Arm (N=131)
MS relapse (Nervous system disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Continuation Arm (N=128) | Drug Discontinuation Arm (N=131)
MS relapse (Nervous system disorders) | 0 (0) | 3 (3)
New MS MRI lesion (Nervous system disorders) | 5 (5) | 14 (16)
Leg edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leptomeningeal enhancement (Nervous system disorders) | 0 (0) | 1 (1)
Elevated PSA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abnormal white blood cell count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abnormal glucose level (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Injection reaction (General disorders) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 3 (3) | 7 (7)
Urinary tract infection (Renal and urinary disorders) | 17 (27) | 11 (26)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 12 (13) | 13 (14)
Influenza (Infections and infestations) | 4 (4) | 10 (10)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 14 (14)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 30 (37)

LIMITATIONS AND CAVEATS:
Mostly white women; all participants in US; Relatively short follow-up (maximum 2 years); Most participants using older, injectable therapies for MS; Small numbers don't allow for significant subgroup analysis, eg not enough on high efficacy medications; Being a pragmatic study (real-world, insurance paid for MRI scans), and COVID pandemic resulted in more missing data than desirable; No brain volume data, a meaningful measure; No NfL or other serum or spinal fluid biomarker data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03073603/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03073603/ICF_001.pdf